CLINICAL TRIAL: NCT02968875
Title: Alzheimer's Disease and Physiological, Cognitive Function and BDNF Levels of Plasma Adaptation After Exercise Training
Acronym: MARAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15/B/03
Record Dates: First submitted 2016-09-07; First posted 2016-11-21 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer's Disease
Keywords: endurance training; BDNF analysis; cognitive function; physiological abilities
MeSH Terms: conditions — Alzheimer Disease | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endurance Training (Active Comparator): The first group of 40 people will do endurance training; 20 of them will perform a continuous exercise on cycle ergometer at a power equivalent to 70% of the maximal heart rate, twice a week. The other group will do Interval Training, with a four minute long base and one minute long peak, twice a week. The base workload will be equivalent to an intensity of 60% of the maximal heart rate and the peak will be equivalent to 80% of the maximal heart rate.
  Interventions: Device: Endurance Training
- Control group (Active Comparator): 20 persons will be in the control group and they will not perform the endurance training. However, they will have 9 therapeutic education meetings.
  Interventions: Other: therapeutic education meetings

INTERVENTIONS:
Device: Endurance Training — 40 people will submitted to endurance training: 20 will perform a continuous training and 20 will perform an interval training. The variables that will be analyzed are maximum aerobic power, endurance, heart rate, prehension strength, Mini-Mental State Examination (MMSE), REY's test, biological examination and level of BDNF plasma, before and after the intervention and one month after the end of the intervention and one month after the end of the intervention.
  Arms: Endurance Training
Other: therapeutic education meetings — Group of 20 people will be the control group and will not perform ET. However, they will have 9 therapeutic education meetings.
  Arms: Control group

SUMMARY:
Alzheimer's disease (AD) is a neurodegenerative disease leading to one of the most common forms of dementia in humans and memory disorder is one of the first symptoms that lead to diagnosis.

DETAILED DESCRIPTION:
Present in greater amounts in the regions of the hippocampus and cortex, the Brain-derived neurotrophic factor (BDNF) is essential to both learning and memory processes. This protein is found in lower amounts in people with AD. Acute physical activity of moderate to vigorous intensity would increase the levels of plasma BDNF whether for a healthy person or a person with AD. Nevertheless in rest, healthy people have higher level of BDNF than individuals with AD. There are no studies on the effect of chronic exercise based on BDNF level at rest in people with AD. In a hypothetical endurance training of 18 sessions, whether interval or continuous training the levels of BDNF would increase in people with AD at rest. Their physiological and neuropsychological performances would also show a rise.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease patients diagnosed by a consultation memory (DSM- IV)
* Person with at least 60 years
* Person with a score higher than 15 in the Mini Mental State Examination
* No one can achieve the pedaling motion
* People who do not perform regular physical activity on bike
* Nobody has given free and informed consent in writing or obtained from a trusted person or the family environment
* People affiliated to a social security

Exclusion Criteria:

* Patient who refused to provide written consent
* Inability to pedal
* Recent myocardial necrosis (less than 3 months)
* Aortic Stenosis
* Uncompensated heart failure
* Unstable angina
* Ventricular arrythmia
* Pulmonary embolism
* Coxarthrosis, knee, ankle osteoarthritis
* Not affiliated to a social security
* Patient already participating in another biomedical research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Measuring the effect of a program of endurance training (ET), on the levels of plasma BDNF. | Up to 4 months

SECONDARY OUTCOMES:
Measuring the effect of training on the psychological performance by using questionnaire MMSE | Up to 4 months
Measuring the effect of training on the psychological performance by using questionnaire: Rey auditory verbal learning test (RAVLT) | Up to 4 months
Measuring the effect of training on the psychological performance by using questionnaire: quality of life (QoL-AD) | Up to 4 months
Stress test | Up to 4 months
  Measuring the effect of training on the physiological performance by determining the maximum power of the effort tolerated
Stress test | Up to 4 months
  Measuring the effect of training on the physiological performance by determining the grip strength
Measuring the effect of training on the physiological performance with a walk test of 6 minutes. | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ms FANON, Doctor, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Enette L, Vogel T, Merle S, Valard-Guiguet AG, Ozier-Lafontaine N, Neviere R, Leuly-Joncart C, Fanon JL, Lang PO. Effect of 9 weeks continuous vs. interval aerobic training on plasma BDNF levels, aerobic fitness, cognitive capacity and quality of life among seniors with mild to moderate Alzheimer's disease: a randomized controlled trial. Eur Rev Aging Phys Act. 2020 Jan 6;17:2. doi: 10.1186/s11556-019-0234-1. eCollection 2020. PMID 31921371